CLINICAL TRIAL: NCT05721040
Title: Short-term Evaluation of Motor and Sensory Function in Post-COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Lecturer of chest diseases and tuberculosis, Assiut University
Other Study IDs: Covid-19 NCS
Record Dates: First submitted 2023-02-07; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Motor Neuropathy; Sensory Neuropathy
Keywords: Covid-19; Nerve conduction studies; Neuropathy; Complication
MeSH Terms: conditions — Neuritis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Group: Motor nerve study was performed in the median and posterior tibial nerve to assess the motor function of the upper and lower limbs.
  Sensory nerve study was done for the median and sural nerves to estimate the peripheral neurological function of both upper and lower limbs.
  F wave study was performed for the upper limb in the median nerve.
- Control Group: Motor nerve study was performed in the median and posterior tibial nerve to assess the motor function of the upper and lower limbs.
  Sensory nerve study was done for the median and sural nerves to estimate the peripheral neurological function of both upper and lower limbs.
  F wave study was performed for the upper limb in the median nerve.

SUMMARY:
SARS-COV-2 infection reframed medical knowledge in many aspects, yet there is still a lot to be discovered. our aim is to evaluate neurological impact of covid-19; if there is any.

DETAILED DESCRIPTION:
Coronavirus disease 19 (COVID-19) can cause neuropsychiatric, psychological and psychosocial impairments. Literature regarding the sensory and motor affection of COVID-19 is still limited.

Public health emergencies as COVID-19 are likely to cause adverse neuropsychiatric impacts. Cognitive impairments after SARS-COV-2 infection were noticed, COVID-19 patients complain of poor concentration, declined memory, and insomnia, as well as anxiety and depression symptoms.

in a study; Neurological manifestations described in 36.4% of 214 patients with confirmed COVID-19. However, the symptoms described [dizziness (not further defined), headache, and impaired consciousness] are commonplace in many severe infections and represent disturbances in neurological function rather than a neurological disease per se. Anosmia and ageusia have received much attention, but are ubiquitous in other common upper respiratory tract infections. While a reported increased risk of cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed RT-PCR COVID-19 infection with mild to moderate severity based on the Egyptian ministry of health (MOH) protocol (version 1.4, November 2020) with neurological symptoms suggestive of peripheral neuropathy

Exclusion Criteria:

* patients presenting with neurological manifestations other than peripheral neuropathy, such as stroke, cerebral hemorrhage, encephalitis, or meningitis.
* Patients with any medical condition or comorbidities that may affect the result of the study as diabetes, arthritis, and carpel tunnel syndrome.
* Severe COVID-19 patients with a critical condition that needs hospitalization and ventilatory support were also excluded from the study.

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 RT-PCR-confirmed COVID-19 patients with neurological manifestations presented at outpatient clinics of chest and neurology departments were recruited. Twenty healthy age and gender-matched volunteers were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Motor nerve function | 1 MONTH
  The motor nerve study was performed in the median and posterior tibial nerve to assess the motor function of the upper and lower limbs; included Compound motor action potential (CMAP), Motor nerve conduction velocity (MNCV), and nerve conduction latency recording.
Sensory nerve function | 1 MONTH
  The sensory nerve study was done for the median and sural nerves including Sensory motor nerve conduction amplitude, latency, and velocity were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Gamal Elddin Khaleel, Lecturer, Principal Investigator — Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Egypt

REFERENCES:
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Elshebawy H, Ezzeldin MY, Elzamarany EH. Characteristics of COVID and post COVID polyneuropathies in adults and pediatrics: an Egyptian sample. Egypt J Neurol Psychiatr Neurosurg. 2021;57(1):178. doi: 10.1186/s41983-021-00435-9. Epub 2021 Dec 20. PMID 34955631
- [Background] Ellul MA, Benjamin L, Singh B, Lant S, Michael BD, Easton A, Kneen R, Defres S, Sejvar J, Solomon T. Neurological associations of COVID-19. Lancet Neurol. 2020 Sep;19(9):767-783. doi: 10.1016/S1474-4422(20)30221-0. Epub 2020 Jul 2. PMID 32622375